CLINICAL TRIAL: NCT07317388
Title: Study on the Effectiveness of Group Psychoeducation (for Users and Caregivers) in Promoting Autonomy at Home for Individuals With Psychatric Disorder.
Brief Title: Group Psychoeducation to Promote Independent Living in Individuals With Psychiatric Disorders
Acronym: AUTON'HOME
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Raluca ROSETTI, Principal Investigator, Centre hospitalier de Ville-Evrard, France
Other Study IDs: 0098_EPSVE_AUTON'HOME
Record Dates: First submitted 2025-09-26; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Psychiatric Disorder
Keywords: psychoeducation; autonomy; mental health; group therapy; independent living
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AUTON'HOME Group 1: Group of 6 patients with severe mental disorders (mood or psychotic disorders), residing in Seine-Saint-Denis, supported by the RPS platform. They participate in a 10-week psychoeducation program called 'AUTON'HOME', aimed at improving their autonomy at home. The program includes 10 thematic sessions on cognitive functions, daily living skills, hygiene, housing management and social participation. Evaluations are conducted before and 3 months after the program.
- AUTON'HOME Group 2: Group of 6 patients with severe mental disorders (mood or psychotic disorders), residing in Seine-Saint-Denis, supported by the RPS platform. They participate in a 10-week psychoeducation program called 'AUTON'HOME', aimed at improving their autonomy at home. The program includes 10 thematic sessions on cognitive functions, daily living skills, hygiene, housing management and social participation. Evaluations are conducted before and 3 months after the program.
- AUTON'HOME Group 3: Group of 6 patients with severe mental disorders (mood or psychotic disorders), residing in Seine-Saint-Denis, supported by the RPS platform. They participate in a 10-week psychoeducation program called 'AUTON'HOME', aimed at improving their autonomy at home. The program includes 10 thematic sessions on cognitive functions, daily living skills, hygiene, housing management and social participation. Evaluations are conducted before and 3 months after the program.
- AUTON'HOME Group 4: Group of 6 patients with severe mental disorders (mood or psychotic disorders), residing in Seine-Saint-Denis, supported by the RPS platform. They participate in a 10-week psychoeducation program called 'AUTON'HOME', aimed at improving their autonomy at home. The program includes 10 thematic sessions on cognitive functions, daily living skills, hygiene, housing management and social participation. Evaluations are conducted before and 3 months after the program.

SUMMARY:
This study evaluates the effectiveness of group psychoeducation for users and carers to help people with severe psychiatric disorders achieve autonomy at home.

DETAILED DESCRIPTION:
The study will assess the autonomy of users with severe psychiatric disorders in a home setting before and after participation in the psychoeducation group. The program includes 10 sessions focusing on various aspects of daily living and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer for a home autonomy project
* Management of a mental health problem (mood disorder or psychotic disorder)
* Consent for participation (non-opposition)
* Taken care by the RPS 93 platform

Exclusion Criteria:

* Acute clinical state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with severe psychiatric disorders, managed by the RPS 93 platform, and volunteers for a home autonomy project.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Life Habits Assessment Tool | Baseline, at the end of the 10-week AUTON'HOME psychoeducation program, and 3 months after program completion
  Assessing the autonomy of users with severe psychic pathologies in housing before and after participation in the psychoeducation group.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale | Baseline, at the end of the 10-week AUTON'HOME psychoeducation program, and 3 months after program completion
  Assesses emotional impressions and depressive symptoms in caregivers.
Zarit Burden Interview Scale | Baseline, at the end of the 10-week AUTON'HOME psychoeducation program, and 3 months after program completion
  Quantifies caregiver burden.
Family Expectations Questionnaire | Baseline (prior to initiation of the AUTON'HOME psychoeducation program)
  It aims to collect the expectations of family members regarding the autonomy and daily functioning of their loved one living with a severe mental disorder.
Family Expectations Fulfillment Questionnaire | At the end of the 10-week AUTON'HOME psychoeducation program and 3 months after program completion
  It evaluates whether the expectations previously expressed by the family have been fulfilled, partially met, or unmet.
Positive and Negative Syndrome Scale | Baseline and 3 months after completion of the 10-week AUTON'HOME psychoeducation program
  Measures severity of psychiatric symptoms.
Clinical Global Impression | Baseline and 3 months after completion of the 10-week AUTON'HOME psychoeducation program
  Assesses global improvement compared to baseline.
Montreal Cognitive Assessment | Baseline and 3 months after completion of the 10-week AUTON'HOME psychoeducation program
  Screens for mild to moderate cognitive impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Raluca ROSETTI, Docrorat d'Etat en Médecine, Principal Investigator — EPS VILLE EVRARD
Locations (1):
- EPS VIlle Evrard - UNIRRE 93, Neuilly-sur-Marne, France

REFERENCES:
- [Result] Xia J, Merinder LB, Belgamwar MR. Psychoeducation for schizophrenia. Cochrane Database Syst Rev. 2011 Jun 15;2011(6):CD002831. doi: 10.1002/14651858.CD002831.pub2. PMID 21678337
- [Result] Somerville, P., (1998). " Empowerment through Residence ", Housing Studies, Vol. 13, n° 2, pp. 233-258.
- [Result] Richard, M.-J., Touroude, R., Loubier , D. (2018) Habitat et accompagnement. Santé mentale, 228, 42-47.
- [Result] Pan AW, Fisher AG. The Assessment of Motor and Process Skills of persons with psychiatric disorders. Am J Occup Ther. 1994 Sep;48(9):775-80. doi: 10.5014/ajot.48.9.775. PMID 7977620
- [Result] Mausbach BT, Bowie CR, Harvey PD, Twamley EW, Goldman SR, Jeste DV, Patterson TL. Usefulness of the UCSD performance-based skills assessment (UPSA) for predicting residential independence in patients with chronic schizophrenia. J Psychiatr Res. 2008 Mar;42(4):320-7. doi: 10.1016/j.jpsychires.2006.12.008. Epub 2007 Feb 15. PMID 17303168
- [Result] Leguay D, Cochet A, Matignon G, Hairy A, Fortassin O, Marion JM. [Social Autonomy Scale. First validation data]. Encephale. 1998 Mar-Apr;24(2):108-19. French. PMID 9622789
- [Result] Latalova K. Insight in bipolar disorder. Psychiatr Q. 2012 Sep;83(3):293-310. doi: 10.1007/s11126-011-9200-4. PMID 22101737
- [Result] Gaudelus, B., (2018). Quels outils pour évaluer la capacité à habiter, Santé mentale, 228,48-54.
- [Result] Beaulieu A, Morin P, Provencher H, Dorvil H. [Work as a social determinant of health for mental health services consumers.]. Sante Ment Que. 2002;27(1):177-93. French. PMID 18253624
- [Result] Chambon, N., Picolet, É. & Sorba, M. (2020). L'intervention sociale à l'épreuve d'une préoccupation pour la santé mentale. Mobilisation du rétablissement et politique de logement d'abord. Revue française des affaires sociales, 97-116.
- [Result] Barres, M., (2016) L'action de la psychiatrie pour l'accès et le maintien dans le logement des personnes vivant avec des troubles psychiques en Île-de-France. https://bibliotheques.ghu-paris.fr/doc_num.php?explnum_id=1299
- [Result] Bond K, Anderson IM. Psychoeducation for relapse prevention in bipolar disorder: a systematic review of efficacy in randomized controlled trials. Bipolar Disord. 2015 Jun;17(4):349-62. doi: 10.1111/bdi.12287. Epub 2015 Jan 16. PMID 25594775
- [Result] Baier M. Insight in schizophrenia: a review. Curr Psychiatry Rep. 2010 Aug;12(4):356-61. doi: 10.1007/s11920-010-0125-7. PMID 20526897
- [Result] Amado, C., Musset, T., & Gozlan, G., (2018). Le SAMSAH'Appart, espace d'évaluation et d'apprentissage. Santé mentale, 228, 69-70.
- [Result] Alhadidi MM, Lim Abdullah K, Yoong TL, Al Hadid L, Danaee M. A systematic review of randomized controlled trials of psychoeducation interventions for patients diagnosed with schizophrenia. Int J Soc Psychiatry. 2020 Sep;66(6):542-552. doi: 10.1177/0020764020919475. Epub 2020 Jun 7. PMID 32507073